CLINICAL TRIAL: NCT04544098
Title: A Pilot Study Investigating Intrahepatic Arterial And Intravenous Infusion Of The Radiolabeled Somatostatin Agonist 177Lu-DOTATATE In Patients With Liver-Dominant Metastatic Gastroenteropancreatic (GEP), Bronchial or Unknown Primary Well Differentiated Neuroendocrine Tumors
Brief Title: Lutathera in People With Gastroenteropancreatic (GEP), Bronchial or Unknown Primary Neuroendocrine Tumors That Have Spread to the Liver
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-232
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Neuroendocrine Tumors; Liver-Dominant Metastatic Pancreatic Neuroendocrine Tumors
Keywords: 177Lu-DOTATATE; Pan-NETs; Intrahepatic Arterial; Intravenous Infusion; Gastroenteropancreatic (GEP),; Bronchial or Unknown Primary Well Differentiated Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — lutetium Lu 177 dotatate

STUDY DESIGN:
Intervention Model Description: This is an early-phase trial in which a total of 10 patients with progressive, inoperable, liver-dominant, metastatic GEP, bronchial or unknown primary NETs will be enrolled in this combined intraarterial/intravenous therapeutic approach with 177Lu-DOTATATE.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PRRT with 177Lu-DOTATATE (Experimental): Patients will undergo a routine 68Ga-DOTATATE PET/CT. Patients with sufficient tumor uptake will be offered therapy with 177Lu-DOTATATE. The treatment regimen will consist of four administrations of 177Lu-DOTATATE-two intra-arterial followed by two intravenous, two months apart (+/- 2 weeks), with renal protective amino acid solution co-administration.
  Interventions: Drug: 177Lu-DOTATATE

INTERVENTIONS:
Drug: 177Lu-DOTATATE — The treatment regimen will consist of four administrations of 177Lu-DOTATATE-two intra-arterial followed by two intravenous, two months apart (+/- 2 weeks), with renal protective amino acid solution co-administration. The activity per cycle will be fixed for each patient: patients will receive two intra-arterial cycles of 7.4 GBq, unless toxicity occurs requiring dose modifications.

SUMMARY:
This study will look at whether it is practical and safe to give Lutathera directly into an artery of the liver (hepatic intraarterial infusion). The researchers will compare the effects of hepatic intraarterial infusion in the liver with the effects of the standard approach (intravenous infusion in the arm). The researchers will also determine whether Lutathera is effective against participants' cancer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects affected by histologically proven, somatostatin-receptor positive, progressive, nonresectable, liver-dominant metastatic GEP, bronchial or unknown primary tumors, G1, G2 and G3, according to the new WHO classification of 2017.

  1. Ability to understand and willingness to sign a written informed consent document
  2. Aged 18 years or older
  3. Histologically proven or cytologically confirmed, non-resectable,GEP, bronchial or unknown primary NETs with liver-dominant disease with or without prior treatment with embolization
  4. Measurable disease as defined by RECIST 1.1 with at least one dimension ≥ 1.0 cm
  5. GEP or unknown primary NET of grade 1, 2 and 3 according to WHO 2017, typical or atypical lung carcinoid according to the Travis classification of 2004
  6. Progression of disease defined by one of the following occurring within 6 months of study entry:

     1. At least a 20% increase in radiologically or clinically measurable disease;
     2. Appearance of any new lesion;
     3. Symptomatic disease (including worsening hormonal symptoms or symptoms related to tumor burden);
  7. Overexpression of somatostatin receptors of the target lesions at 68Ga-DOTATATE PET/CT with SUV of lesions greater than normal liver at least in 1 metastasis.
  8. ECOG performance status 0 or 1 (Karnofsky ≥ 70%).
  9. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
  10. Previous local therapy (e.g., chemoembolization or bland embolization) is allowed if completed >6 weeks prior to study entry. For such patients, there must be either progression of measurable disease documented within the treatment field, or measurable progressive disease outside the treatment field prior to study entry.
  11. Previous oral chemotherapy, biotherapy (such as Interferons or Everolimus) and/or investigational agents are allowed if completed >4 weeks prior to study entry For patients who received systemic therapy prior to study entry, there must be documented progression of measurable disease since receiving systemic therapy prior to study entry.
  12. Patients must not be candidate for potentially curative surgery. Prior surgery is allowed no less than 6 weeks prior to study entry. Note: Patients who have disease that is amendable to resection but who are not a surgical candidate for other medical reasons would be permitted.

Exclusion Criteria:

1. Women who are pregnant or breastfeeding
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-DOTATATE as assessed from medical records.
3. Life expectancy < 6 months as assessed by the treating physician.
4. Over 80% liver involvement by tumor per the judgement of the radiologist
5. Poorly differentiated neuroendocrine neoplasms (Neuroendocrine Carcinoma), small and large cell type; Mixed Neuroendocrine-Nonneuroendocrine Neoplasm (MiNEN).
6. Presence of somatostatin receptor negative lesions.
7. Prior treatment with other radiolabeled somatostatin analogs.
8. Prior systemic chemotherapy, except oral chemotherapy with capecitabine + temozolomide
9. Contraindication to angiography/embolization including:

   1. Patients cannot receive contrast
   2. Severe allergic reaction to contrast despite premedication. Patients in who IV contrast is contraindicated are recommended to have MRI abdomen and noncontrast chest CT scan.
   3. Poor renal function not on dialysis
   4. Other, based on judgment of the investigator
10. Main portal vein tumor thrombus.
11. Deteriorated renal function:

    1. Serum creatinine >1.7 mg/dL OR
    2. EGFR <30 ml/min
12. Deteriorated bone marrow function:

    1. Hb <8.0 g/dL;
    2. WBC <3000/mm3;
    3. ANC<1500/mm3;
    4. Platelets <75.000/mm3
13. Deteriorated liver function:

    1. INR > 2.0 for patients that are not on Coumadin or Xarelto
    2. PTT > 2x ULN
    3. Total bilirubin >3 mg/dl
    4. Serum albumin <3.0 g/dL unless prothrombin time is within the normal range.
14. Clinically relevant toxicities from prior therapies that have not resolved to grade 1 or grade 0
15. Previous liver radioembolization with 90Y-microspheres.
16. Known brain metastases and/or carcinomatous meningitis, unless these metastases have been treated and stabilized.
17. Uncontrolled diabetes mellitus
18. Inability to interrupt short-acting Octreotide for 24 h before and 24 h after the administration of 177Lu-DOTATATE; inability to have an interval between Octreotide LAR and 177Lu-DOTATATE of ≥4 weeks
19. Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
20. Prior external beam radiation therapy involving >25% of the bone marrow.
21. Unmanageable urinary incontinence rendering the administration of 177Lu-DOTATATE unsafe
22. Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and with no evidence of recurrence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
number of patients who successfully complete 2 IA injections | 2 years
  Feasibility will be defined as at least 7 or more patients out of 10 patients who successfully complete 2 IA injections.
Objective response | 1 year
  classified according to RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bodei, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm